CLINICAL TRIAL: NCT03955055
Title: A Randomized Comparison of Early Deployment of a Video Capsule (Endocapsule EC-10: Olympus Tokyo) in Clinical Decision Unit (CDU) Versus Standard of Care (SOC) Work-up of Hematemesis [H] and Non-hematemesis Gastrointestinal Bleeding [NHGIB]
Brief Title: Study of Early Endocapsule (EC) in Clinical Decision Unit Versus Standard of Care Work-up for GI Bleeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christopher Marshall (Other)
Collaborators: Olympus Corporation of the Americas (Industry)
Responsible Party: Sponsor-Investigator, Christopher Marshall, Assistant Professor of Medicine, University of Massachusetts, Worcester
Organization: University of Massachusetts, Worcester (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: H00015196
Record Dates: First submitted 2019-05-16; First posted 2019-05-17 (Actual); Results first posted 2023-07-10 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Gastro Intestinal Bleeding; Hematemesis; Melena
Keywords: Gastro Intestinal Bleeding
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Hematemesis; Melena | interventions — Capsule Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Early Capsule Group (Experimental): The intervention for subjects in this arm will be to have a video capsule deployed as soon as possible after presentation to the clinical decision unit. Information from the video capsule will be obtained and reviewed to determine location of bleeding. Once that information has been obtained a decision will be made on which endoscopic test is most pertinent in finding and treating the source of bleeding.
  Interventions: Device: Video Capsule Endoscopy
- Standard of Care Work-up (No Intervention): In this arm, patients will receive "standard of care workup" for non-hematemesis gastrointestinal bleeding. This could include upper endoscopy, colonoscopy, and additional capsule or small bowel enteroscopy depending on the subject's presentation and the results of the workup performed by the gastroenterology team. For patients requiring a video capsule endoscopy as part of "standard of care workup" the patients will be given the same Olympus video capsule that is used in the "Early Capsule" group.

INTERVENTIONS:
Device: Video Capsule Endoscopy — Patients will swallow a video capsule as soon as possible (immediately or within 10 hours, if patient is not fasting).
  Other Names: Olympus EndoCapsule EC-10
  Arms: Early Capsule Group

SUMMARY:
This study will evaluate the use of the Olympus EndoCapsule EC-10 video capsule compared with the standard of care workup for patients in the Clinical Decision Unit who have symptoms of gastrointestinal (GI) bleeding. Patients will be eligible if they have any symptoms of GI bleeding, either vomiting blood or symptoms without vomiting blood.

Patients randomized to the early capsule arm will have an immediate video capsule endoscopy. Patients randomized to the standard of care arm will have no study intervention and will follow the treating physician's diagnostic workup.

The primary goal of the study is to compare how often a source of bleeding is identified in patients in the two groups.

DETAILED DESCRIPTION:
After 40 years of considering gastrointestinal bleeding as upper or lower and largely ignoring the small intestine, there is accumulating evidence that the conventional approach to the assessment of non-hematemesis gastrointestinal bleeding (NHGIB) could be improved by early deployment of a video capsule as the first diagnostic test. Currently, video capsule endoscopy (VCE) is considered the gold standard diagnostic test for small intestinal bleeding after upper and lower endoscopy. However, video capsule endoscopy is an underutilized, minimally invasive tool that can improve rates of detection, minimize patient discomfort, and shorten the length of hospital stay for many patients. In a recent study at University of Massachusetts Worcester (UMass) of 336 patients who presented to the Emergency Department (ED) with complaints of gastrointestinal bleeding only 36 patients (10.7%) were given a video capsule during their stay.1

Traditionally, in patients with hematemesis (H), upper endoscopy has been the diagnostic and therapeutic modality of choice. However, recent data from a randomized clinical trial suggests that when video capsule endoscopy is used as the primary diagnostic tool, the investigators were able to safely define those patients that require admission from those that can be discharged for later follow-up 2. In this cohort, 30% of patients could be safely discharged and undergo endoscopy, if necessary within 48 hours, as an outpatient. This data is consistent with internal epidemiological data from UMass where nearly 30% of patients who were admitted did not receive any endoscopic evaluation as in-patients.

Similarly, a randomized controlled trial has recently shown that patients with NHGIB may benefit from early VCE. In this population, the detection of active bleeding with video capsule as the first procedure was 63% compared with 27% for the standard of care approach. The study did not demonstrate a significant reduction in length stay since this was not part of the trial design. No attempt was made to change physician behavior. The study was too small to demonstrate a reduction in procedures, but there was a modest reduction in healthcare costs despite the addition of the video capsule. The study encountered no adverse events. Readmission rates were not significantly reduced but there were no re-admissions in the capsule group for gastrointestinal (GI) bleeding where there were four in the standard of care group.

The hypothesis is that both signs and symptoms provide poor localization as to the origin of bleeding in NHGIB. Data from the previous study suggests that the ingestion of a video capsule in the emergency department could quickly and non-invasively provide clinicians accurate data as to the origin of the bleeding. This information could provide a guide to further management of the patient. Video capsule endoscopy is able to visualize bleeding in the esophagus, stomach, duodenum, small intestine and right colon, thereby eliminating the guess work of deciding which endoscopic approach to use.

The study plans to use the clinical decision unit for two reasons. This unit provides an ideal site for the early safe deployment of a video capsule or initiation of a standard of care workup for either or NHGIB. Second, in those patients who are demonstrated not to be bleeding in either group by capsule endoscopy or standard of care workup may be discharged home safely without being admitted, thereby saving significant costs. It is known that 80% of patients stop bleeding spontaneously. Thus, the earlier they are examined the more likely the origin of the bleeding is likely to be found and appropriate management instituted.

The use of capsule endoscopy has been approved by the FDA since 2001 for small intestinal bleeding obscure GI Bleeding. It is very safe, no deaths associated with its use have been reported. More than 3 million capsules have been deployed and obstruction and perforation are extremely rare.

Interest in the broader use of VCE is accumulating. A pilot study on the use of early use of VCE in acute NHGIB showed a 50% reduction to time to diagnosis in 24 patients. More recently studies of VCE deployed in the ED, in patients with upper GI bleeding showed improved management. The UMass group recently demonstrated that the closer a video capsule is performed to the time of bleeding the higher the likelihood of locating the sources and the higher the therapeutic intervention rate.

This protocol is logical step to prospectively examine this concept in a large randomized prospective trial for both H and NHGIB. The questions are, can early capsule intervention decrease time to diagnosis, numbers of procedures, admission rate and hospital length of stay in patients with H and NHGIB.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years old
* New onset of hematemesis, melena or hematochezia
* Able to sign consent
* Hemodynamically stable (that is, blood pressure >100/60 or pulse <110 at the time of consent)
* Emergency Department must plan to admit patient to the hospital or Clinical Decision Unit
* If patients have pacemakers and/or implantable cardioverter defibrillator (ICD), they will be placed on telemetry

Exclusion Criteria:

* adults unable to consent
* individuals who are not yet adults (infants, children, teenagers)
* pregnant women
* prisoners
* prior history of gastroparesis
* prior history of gastric or small bowel surgery
* prior history of inflammatory bowel disease
* concern for infectious colitis
* evidence of dysphagia at the time of presentation
* presence of small amounts of bright red blood per rectum
* allergy to metoclopramide or erythromycin
* code status of do not resuscitate/do not intubate (DNR/DNI) or comfort measures only (CMO)
* prior history of abdominal radiation
* abdominal pain suggesting an acute abdomen or obstruction.
* patients who cannot undergo surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2020-02-04 (Actual); Primary Completion 2022-04-09 (Actual); Study Completion 2022-04-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Marshall, MD, Principal Investigator — UMass Medical School Assistant Professor of Medicine
Locations (1):
- UMass Memorial Medical Center, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marya NB, Jawaid S, Foley A, Han S, Patel K, Maranda L, Kaufman D, Bhattacharya K, Marshall C, Tennyson J, Cave DR. A randomized controlled trial comparing efficacy of early video capsule endoscopy with standard of care in the approach to nonhematemesis GI bleeding (with videos). Gastrointest Endosc. 2019 Jan;89(1):33-43.e4. doi: 10.1016/j.gie.2018.06.016. Epub 2018 Jun 20. PMID 29935143
- [Background] Singh A, Marshall C, Chaudhuri B, Okoli C, Foley A, Person SD, Bhattacharya K, Cave DR. Timing of video capsule endoscopy relative to overt obscure GI bleeding: implications from a retrospective study. Gastrointest Endosc. 2013 May;77(5):761-6. doi: 10.1016/j.gie.2012.11.041. Epub 2013 Feb 1. PMID 23375526
- [Background] Jawaid S, Gondal B, Singh, A, Marshall C, and Cave D. The epidemiology of gastrointestinal bleeding in an academic emergency department as a basis for reconfiguring the conventional approach to its diagnosis and management. Gastrointestinal Endoscopy 2013;77:Supplement, Page AB483.
- [Background] Jawaid S, Marya N, Gondal B, Maranda L, Marshall C, Charpentier J, Singh A, Foley A, and Cave D. . A reconsideration of the diagnosis and management of gastrointestinal bleeding based on its epidemiology and outcomes analysis. Gastrointestinal Endoscopy 2014;79:Supplement, Page AB231.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Early Capsule Group | Standard of Care Work-up
Started | 15 | 20
Completed | 14 | 18
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Early Capsule Group | Standard of Care Work-up | Total
Number analyzed (Participants) | 15 | 20 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.47 (11.27) | 66.45 (16.09) | 65.17 (14.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 12 | 14 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 14 | 20 | 34
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 13 | 18 | 31
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Rate of Detection of Bleeding
Description: Rate of detection of active bleeding or stigmata of recent bleeding [blood clot or visible vessel]
Time Frame: Enrollment to time of detection of bleeding as measured in hours, up to 720 hours, whichever is sooner
Population: One participant excluded, unable to swallow capsule
Measure: Count of Participants; unit: Participants
Arm/Group | Early Capsule Group | Standard of Care Work-up
Number analyzed (Participants) | 14 | 20
Participants | 11 | 11

2. Primary Outcome: Time to Detection of Bleeding
Description: Time to detection of active bleeding or stigmata of recent bleeding [blood clot or visible vessel]
Time Frame: Enrollment to time of detection of bleeding as measured in hours, up to 720 hours, whichever is sooner
Population: Time point data was missing on several participants.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Early Capsule Group | Standard of Care Work-up
Number analyzed (Participants) | 3 | 6
hours | 20.9 (1.9) | 17.7 (9.5)

3. Secondary Outcome: Admission Rate
Description: Rate of in-patient admissions to the hospital
Time Frame: Enrollment to time of admission as measured in hours, up to 720 hours, whichever is sooner
Population: One participant was excluded due to inability to swallow capsule.
Measure: Count of Participants; unit: Participants
Arm/Group | Early Capsule Group | Standard of Care Work-up
Number analyzed (Participants) | 14 | 20
Participants | 14 | 20

4. Secondary Outcome: Re-admission Rate
Description: Rate of in-patient re-admissions to the hospital
Time Frame: Enrollment to 720 hours
Population: One participant was excluded due to inability to swallow capsule.
Measure: Count of Participants; unit: Participants
Arm/Group | Early Capsule Group | Standard of Care Work-up
Number analyzed (Participants) | 14 | 20
Participants | 4 | 2

5. Secondary Outcome: Hospital Length of Stay
Description: Length of hospital stay measured in hours
Time Frame: Enrollment to time of discharge as measured in hours, up to 720 hours, whichever is sooner
Population: One participant excluded due to inability to swallow capsule.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Early Capsule Group | Standard of Care Work-up
Number analyzed (Participants) | 14 | 20
hours | 143.7 (102.3) | 140.9 (80.5)

6. Secondary Outcome: Endoscopic Procedures
Description: Number of endoscopic procedures performed
Time Frame: Enrollment to 720 hours
Population: One participant excluded due to inability to swallow capsule.
Measure: Mean (Standard Deviation); unit: procedures
Arm/Group | Early Capsule Group | Standard of Care Work-up
Number analyzed (Participants) | 14 | 20
procedures | 1.9 (0.66) | 1.35 (0.67)

7. Secondary Outcome: Therapeutic Procedures
Description: Number of therapeutic procedures performed
Time Frame: Enrollment to 720 hours
Measure: Mean (Standard Deviation); unit: procedures
Arm/Group | Early Capsule Group | Standard of Care Work-up
Number analyzed (Participants) | 14 | 20
procedures | 0.29 (0.47) | 0.35 (0.59)

8. Other Pre Specified Outcome: Complication Rates
Description: Percentage of participants who experienced a complication.
Time Frame: Enrollment to 720 hours
Population: One participant excluded inability to swallow capsule.
Measure: Count of Participants; unit: Participants
Arm/Group | Early Capsule Group | Standard of Care Work-up
Number analyzed (Participants) | 14 | 20
Participants | 6 | 4

9. Other Pre Specified Outcome: Blood Product Transfusions
Description: Number of blood products transfused
Time Frame: Enrollment to one year
Measure: Mean (Standard Deviation); unit: units of packed red blood cells
Arm/Group | Early Capsule Group | Standard of Care Work-up
Number analyzed (Participants) | 15 | 20
units of packed red blood cells | 1.8 (1.6) | 2.2 (2.7)

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Early Capsule Group | Standard of Care Work-up
All-Cause Mortality (participants affected / at risk) | 0/14 | 2/20
Serious Adverse Events (participants affected / at risk) | 4/14 | 3/20
Other Adverse Events (participants affected / at risk) | 1/14 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Early Capsule Group (N=14) | Standard of Care Work-up (N=20)
Melena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Gastrointestinal Bleeding (Gastrointestinal disorders) | 1 (1) | 1 (1)
Hypoxemia (Cardiac disorders) | 0 (0) | 1 (1)
Acute allergic reaction (Immune system disorders) | 1 (1) | 0 (0)
Coronavirus (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Early Capsule Group (N=14) | Standard of Care Work-up (N=20)
Capsule retention (Gastrointestinal disorders) | 1 (1) | 0 (0) — Capsule endoscope was retained, but spontaneously resolved.

LIMITATIONS AND CAVEATS:
The trial was designed before the coronavirus pandemic began and several aspects of the trial were significantly impacted due to the pandemic. The Clinical Decision Unit was effectively closed and endoscopic procedures were limited. While we increased some enrollment in 2021, we were not able to meet our goals due to these unexpected constraints.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2019-05-15): https://cdn.clinicaltrials.gov/large-docs/55/NCT03955055/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-15): https://cdn.clinicaltrials.gov/large-docs/55/NCT03955055/SAP_001.pdf
  • Informed Consent Form (2019-06-06): https://cdn.clinicaltrials.gov/large-docs/55/NCT03955055/ICF_002.pdf